CLINICAL TRIAL: NCT06518187
Title: Investigating the Influence of Catheter Advancement Techniques on Needle Tip Movement During Intravenous Insertion
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202400590
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Health Care Utilization
Keywords: IV Technique
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anesthesiology Healthcare providers/professionals: Investigating whether needle tip movement during catheter advancement is affected by whether the individual performing the insertion pushes the catheter off the needle themselves (either one handed or two handed) or if the catheter is advanced off the needle by another person.
  Interventions: Other: Assessing the impact of three different catheter advancement techniques on needle tip movement during intravenous insertion

INTERVENTIONS:
Other: Assessing the impact of three different catheter advancement techniques on needle tip movement during intravenous insertion — Each participant will perform 3 simulated IV catheter insertions using each of the specified techniques. Participants will use the instrumented 16ga IV catheter to insert into the peripheral vascular access simulator. Needle tip movement (from intent of catheter advancement to 5mm of advancement off the needle) will be measured with 0.2mm accuracy using the electromagnetic tracking technology of the simulator. Data collected will include needle movement after simulated vein punction and during initial catheter advancement off the needle (in mm) which will be recorded within the simulation program and output as a de-identified Excel file

SUMMARY:
This proposed study aims to fill this gap by investigating whether needle tip movement during catheter advancement is affected by whether the individual performing the insertion pushes the catheter off the needle themselves or if it is done by another person.

DETAILED DESCRIPTION:
Participant arrives at the simulation setting. Participant undergoes orientation and consent. This includes orientation to study procedure and equipment, explanation of catheter advancement techniques, and informed consent process. Following consent, participant fills out Participant Questionnaire. Total time required: Approximately 10 minutes.

Participant performs IV catheter insertion using 3 techniques: 1 (Self-advancement single hand), technique 2 (Self-advancement both hands), and technique 3 (second person assisted) in randomized order. Total time required: Approximately 5 minutes. Participant completes Participant Questionnaire. Participant's participation is concluded.

In this study, the observation to be carried out is the total distance of needle tip movement while performing the initial intravenous catheter advancement off of the needle using three different catheter advancement techniques including: Self-advancement with one hand; Self-advancement with two hands; Catheter advancement by another individual.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Willing to consent to the study
3. has some experience placing IV catheters

Exclusion Criteria:

1. Subject refuses to consent
2. Younger than 18 years of age
3. No experience inserting IV catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants for this study are Anesthesiology healthcare professionals/providers who perform IV catheter placement
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Needle tip movement (displacement) in mm during initial advancement of a 16ga IV catheter off of its needle during simulated intravenous catheter insertion with three different catheter advancement techniques.. | 15 minutes
  If there is a significant difference in needle tip movement during catheter advancement related to technique of advancement (one handed, two handed, two person) a preferred technique(s) can be identified

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Gravenstein, MD, Principal Investigator — University of Florida Department of Aneshtesiology
Locations (1):
- UF Health Shands, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT06518187/Prot_SAP_000.pdf